CLINICAL TRIAL: NCT02592018
Title: Characterization of the Response to Secukinumab in Plaque Psoriasis Using Novel Immunologic and Genetic Profiling
Brief Title: Immunologic Response to Secukinumab in Plaque Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CAIN457AUS04T
Record Dates: First submitted 2015-10-16; First posted 2015-10-30 (Estimated); Results first posted 2020-08-27 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Secukinumab (Experimental): All subjects will receive Secukinumab 300mg SQ at weeks 0, 1, 2, 3, 4, and every 4 weeks thereafter until week 48.
  Interventions: Drug: Secukinumab

INTERVENTIONS:
Drug: Secukinumab — Secukinumab 300mg SQ at weeks 0, 1, 2, 3, 4, and every 4 weeks thereafter until week 48. Skin biopsy procedures will be performed at weeks 0, 2, 4, and 12.
  Other Names: Cosentyx

SUMMARY:
This is a single-arm, open-label study, which will examine the effect of secukinumab on the immunologic and genetic environment within psoriatic lesions.

DETAILED DESCRIPTION:
Quantitative analysis of the immunologic changes in immune cell populations will be performed after secukinumab treatment in 15 patients at weeks 2, 4, and 12 compared to baseline week 0. The immunologic profiles in psoriasis patients will also be compared to healthy control skin surgical discard specimens (n=10). The number of differentially expressed genes in each cell population will be quantified by RNA-seq at weeks 2, 4, 12 after secukinumab compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent and comply with the protocol.
2. At least 18 years of age.
3. Diagnosis of predominately plaque psoriasis for at least 6 months prior to enrollment.
4. Subject is considered a candidate for phototherapy or systemic therapy
5. PASI ≥ 12
6. PGA ≥ 3
7. Subject has a negative Quantiferon Gold, or if positive undergoes CXR. If CXR negative, subject initiated prophylactic therapy with isoniazid for a course of 9 months with one month of therapy completed prior to first dose of secukinumab.
8. Subject is unlikely to conceive (male, post-menopausal, or using adequate oral contraceptive therapy or IUD).
9. Physical exam within clinically acceptable limits.

Exclusion Criteria:

1. Subject is unable to provide written informed consent or comply with the protocol.
2. Subject is younger than 18 years of age.
3. Subject has predominately non-plaque form of psoriasis.
4. Subject with mild psoriasis (PASI<12 and PGA<3) or is not a candidate for phototherapy or systemic treatments.
5. Subject has drug-induced psoriasis.
6. Subject with current, or a history of, severe psoriatic arthritis well controlled on current therapy.
7. Subjects with a serum creatinine level exceeding 176.8 μmol/L (2.0 mg/dl).
8. Screening total white blood cell (WBC count) < 2,500/μl, platelets < 100,000/μl, neutrophils < 1,500/μl, or hemoglobin <8.5 g/dl.
9. Evidence of active tuberculosis infection as defined by a positive QuantiFERON TB-Gold test (QFT) with a positive chest X-ray at screening, or untreated latent tuberculosis defined by positive QFT with a negative chest X-ray without prophylactic therapy with isoniazid for a course of 9 months with one month of therapy completed prior to first dose of secukinumab.
10. History of an ongoing, chronic or recurrent infectious disease including past medical history record of HIV, hepatitis B or hepatitis C.
11. Subjects possess other diagnoses that, in the investigator's opinion, preclude him/her from safely participating in this study or interfere with the evaluation of the subject's psoriasis.
12. History of known or suspected intolerance to any of the ingredients of the investigational study product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Liao, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Psoriasis and Skin Treatment Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Secukinumab
Started | 15
Completed | 13
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Secukinumab
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 37 [29 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/Pacific Islander | 4
  Black/African American | 2
  Caucasian | 5
  Hispanic | 4
Family history of psoriasis [Count of Participants; unit: Participants] | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Percentage of CD4+ T Effector Cells Expressing IL17 Compared to Baseline
Time Frame: Baseline to Week 2
Measure: Mean (Standard Deviation); unit: percent change from week 0
Arm/Group | Secukinumab
Number analyzed (Participants) | 15
percent change from week 0 | -1.42 (4.36)

2. Primary Outcome: Change in Percentage of CD4+ T Effector Cells Expressing IL17 Compared to Baseline
Time Frame: Baseline to Week 4
Measure: Mean (Standard Deviation); unit: percent change from week 0
Arm/Group | Secukinumab
Number analyzed (Participants) | 15
percent change from week 0 | 0.23 (8.76)

3. Primary Outcome: Change in Percentage of CD4+ T Effector Cells Expressing IL17 Compared to Baseline
Time Frame: Baseline to Week 12
Measure: Mean (Standard Deviation); unit: percent change from week 0
Arm/Group | Secukinumab
Number analyzed (Participants) | 15
percent change from week 0 | -0.17 (8.73)

4. Secondary Outcome: Change in Number of Differentially Expressed Genes in CD4+ Effectors Compared to Baseline Across All Participants
Description: by RNA-seq
Time Frame: Baseline to Week 2
Measure: Number; unit: genes
Arm/Group | Secukinumab
Number analyzed (Participants) | 15
genes | 67

5. Secondary Outcome: Change in Number of Differentially Expressed Genes in CD4+ Effectors Compared to Baseline
Description: by RNA-seq
Time Frame: Baseline to Week 4
Measure: Number; unit: number of genes
Arm/Group | Secukinumab
Number analyzed (Participants) | 15
number of genes | 308

6. Secondary Outcome: Change in Number of Differentially Expressed Genes in CD4+ Effectors Compared to Baseline
Description: by RNA-seq
Time Frame: Baseline to Week 12
Measure: Number; unit: number of genes
Arm/Group | Secukinumab
Number analyzed (Participants) | 15
number of genes | 1618

7. Secondary Outcome: Change in Number of Differentially Expressed Genes in CD4+ T Regs Compared to Baseline
Description: by RNA-seq
Time Frame: Baseline to Week 2
Measure: Number; unit: number of genes
Arm/Group | Secukinumab
Number analyzed (Participants) | 15
number of genes | 453

8. Secondary Outcome: Change in Number of Differentially Expressed Genes in CD4+ T Regs Compared to Baseline
Description: by RNA-seq
Time Frame: Baseline to Week 4
Measure: Number; unit: number of genes
Arm/Group | Secukinumab
Number analyzed (Participants) | 15
number of genes | 240

9. Secondary Outcome: Change in Number of Differentially Expressed Genes in CD4+ T Regs Compared to Baseline
Description: by RNA-seq
Time Frame: Baseline to Week 12
Measure: Number; unit: number of genes
Arm/Group | Secukinumab
Number analyzed (Participants) | 15
number of genes | 127

10. Secondary Outcome: Change in Number of Differentially Expressed Genes in CD8+ T Effectors Compared to Baseline
Description: by RNA-seq
Time Frame: Baseline to Week 2
Measure: Number; unit: number of genes
Arm/Group | Secukinumab
Number analyzed (Participants) | 15
number of genes | 20

11. Secondary Outcome: Change in Number of Differentially Expressed Genes in CD8+ T Effectors Compared to Baseline
Description: by RNA-seq
Time Frame: Baseline to Week 4
Measure: Number; unit: number of genes
Arm/Group | Secukinumab
Number analyzed (Participants) | 15
number of genes | 102

12. Secondary Outcome: Change in Number of Differentially Expressed Genes in CD8+ T Effectors Compared to Baseline
Description: by RNA-seq
Time Frame: Baseline to Week 12
Measure: Number; unit: number of genes
Arm/Group | Secukinumab
Number analyzed (Participants) | 15
number of genes | 104

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Secukinumab
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab (N=15)
Bell's palsy (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab (N=15)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 2
Upper respiratory infection (Infections and infestations) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-14): https://cdn.clinicaltrials.gov/large-docs/18/NCT02592018/Prot_SAP_000.pdf